CLINICAL TRIAL: NCT01469975
Title: First in Man Study Investigating the Biodistribution, the Safety and Optimal Recommended Dose of a New Radiolabelled Monoclonal Antibody Targeting Frizzled Homolog 10 (FZD10) in Patients With Relapsed or Refractory Non Resectable Synovial Sarcomas
Brief Title: First in Man Study Investigating the Biodistribution, the Safety and Optimal Recommended Dose of a New Radiolabelled Monoclonal Antibody Targeting Frizzled Homolog 10
Acronym: SYNFRIZZ
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Too slow accrual.
Sponsor: Centre Leon Berard (Other)
Collaborators: OncoTherapy Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYNFRIZZ; 2011-002574-23 (EudraCT Number); ET11-062 (Other: Sponsor number)
Record Dates: First submitted 2011-11-03; First posted 2011-11-10 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Sarcoma, Synovial
Keywords: cancer; relapse or refractory
MeSH Terms: conditions — Sarcoma, Synovial; Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: Dose level 1 (Experimental): 1.5 mg of OTSA101-DTPA radiolabelled with 370MBq of 90Y
  Interventions: Drug: OTSA101-DTPA-90Y level 1
- Arm B: Dose level 2 (Experimental): 1.5 mg of OTSA101-DTPA radiolabelled with 1110 MBq of 90Y
  Interventions: Drug: OTSA101-DTPA-90Y level 2
- Arm C: Dose level 3 (Experimental): 3 mg of OTSA101-DTPA radiolabelled with 2220 MBq of 90Y
  Interventions: Drug: OTSA101-DTPA-90Y level 3

INTERVENTIONS:
Drug: OTSA101-DTPA-90Y level 1 — Part 2 of the study 1.5 mg of OTSA101-DTPA radiolabelled with 370MBq of 90Y will be administered IV as a single injection on Day 0.
  Arms: Arm A: Dose level 1
Drug: OTSA101-DTPA-90Y level 2 — Part 2 of the study 1.5 mg of OTSA101-DTPA radiolabelled with 1110 MBq of 90Y will be administered IV as a single injection on Day 0.
  Arms: Arm B: Dose level 2
Drug: OTSA101-DTPA-90Y level 3 — Part 2 of the study 3 mg of OTSA101-DTPA radiolabelled with 2220 MBq of 90Y will be administered IV as a single injection on Day 0.
  This third dose level evaluation will be based on safety and preliminary efficacy data.
  Arms: Arm C: Dose level 3

SUMMARY:
Advanced synovial sarcoma represents an unmet medical need. The gene encoding frizzled homologue 10 (FZD10), a 7-transmenbrane receptor, member of the Wnt signalling receptor family, is overexpressed in SS and is undetectable in normal human tissues except placenta.

OncoTherapy Science Inc. has developed a chimeric humanized monoclonal antibody (mAb) against FZD10, named OTSA101. Non-radiolabeled OTSA101 antibody has only weak antagonistic activity on SS cell growth. However, Yttrium 90-radiolabeled OTSA101 (OTSA101-DTPA-90Y) showed significant antitumor activity following a single intravenous injection in mouse xenograft model.

This first in man clinical trial (Phase I) in relapsing SS patients resistant to Doxorubicin and ifosfamide will be divided in 2 parts.

In Part 1 (imaging part using OTSA101 radiolabelled with Indium 111 [111In]), the biodistribution and tumor uptake of OTSA101-DTPA-111In will be followed using 111In as radiotracer.

In Part 2 (therapeutic part with OTSA101 radiolabelled with Yttrium 90 [90Y]), the safety and PK profiles of OTSA101-DTPA-90Y will be determined and preliminary efficacy data will be collected.

This first in Man study should allow defining the optimal recommended dose of OTSA101-DTPA-90Y.

Patients will be followed during 1 year.

DETAILED DESCRIPTION:
PART 1: Imaging with OTSA101 DTPA-111In OTSA101-DTPA-111In (1.5mg OTSA101-DTPA radiolabeled with 185 MBq of 11In) will be administered intravenously (IV) as a single injection on Day -28 (D-28). Patients will undergo serial anterior-posterior gamma scans and single photon emission computed tomography (SPECT/CT) at 1, 5, 24, 48, 72, 144 hours post-dosing to estimate absorbed radiation doses to tumor, to normal organs (i.e., liver, lung, kidney, and bone marrow), and whole body in order to determine OTSA101-DTPA-111In tumor uptake (ID%/g [% of injected dose (ID) per gram of tumor]) and biodistribution (ratio tumor/normal tissue of estimated radiation-absorbed dose). PK sampling will be performed at the same time points with additional sampling at D-14 and D0.

A Steering Committee meeting is planned at the end of PART 1 for each patient. The Steering Committee will evaluate on a case by case basis at Day -7 for each patient if he/she can proceed to the therapeutic part based on tumor targeting, biodistribution, safety and clinical assessments:

* Patients with expected biodistribution and tumor uptake, no safety concerns and no overt signs of disease progression will proceed to the therapeutic part of the study after validation by the Steering Committee.
* Patients displaying abnormal/unexpected biodistribution of OTSA101-DTPA-111In, safety concerns and/or overt sign of disease progression will be taken off the study and other therapeutic plan will be envisaged.

PART 2: Therapeutic dose of OTSA101-DTPA-90Y OTSA101-DTPA-90Y will be administered IV as a single injection on Day 0 (i.e. 14 days after the injection of OTSA101-DTPA-111In - A 1week-delay [i.e. +7 days] is authorized from the planned D0).

Twelve (12) patients should be randomized in the PART 2 and treated with OTSA101-DTPA-90Y at two initial dose levels (6 patients per dose level):

* Arm A: 1.5 mg of OTSA101-DTPA radiolabeled with 370MBq of 90Y (Dose level 1 (DL1)
* Arm B: 1.5 mg of OTSA101-DTPA radiolabeled with 1110 MBq of 90Y (Dose level 2 (DL2)

Based on safety and preliminary efficacy data, a third dose level will be evaluated in 6 additional patients:

* Arm C: 3 mg of OTSA101-DTPA radiolabeled with 2220 MBq of 90Y (Dose level 3 (DL3).

Such a study design will allow the determination of an optimal and recommended dose, surrounded by a lower suboptimal dose and a higher maximal tolerated (or possibly toxic) dose.

The first 3 patients will be enrolled at Centre Léon Bérard. Following the randomization of the first 2 patients, the accrual will be stopped for a maximal period of 1 month. The safety data will be reviewed every 2 randomized patients. Thee benefit/risk ratio will be regularly reviewed by the iDSMB and the Steering Committee (See Section Study Committee).

A compassionate program is planned for all randomized patients who derive clinical benefit from the study drug (at least stable disease and acceptable tolerance). A maximum of 4 injections per year will be planned. Subsequent injection will be performed provided that the eligibility criteria (except criteria related to previous treatment) are met before the day of administration. All inclusion in the compassionate program will be validated by the Steering Committee.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age ≥ 18 years.
* Histologically confirmed progressive synovial sarcoma with a minimal total tumor volume of 65mL at the time of inclusion.
* Frozen or paraffin-embedded tumor samples for immunohistochemical analysis are mandatory for registration in this study.
* Patients with doxorubicin- and ifosfamide-resistant synovial sarcoma (defined as patients with progression under doxorubicin and ifosfamide treatments or with rapid progression (i.e. within 4 months) after the last dose of doxorubicin and ifosfamide, or patients previously treated with doxorubicin and ifosfamide and with disease progression on another regimen of chemotherapy for advanced disease).
* Patients must have disease not amenable to surgery, radiation or combined modality treatment with curative intent.
* At least one measurable site of disease as defined by RECIST criteria 1.1.
* ECOG performance status of 0, 1, 2.
* Life expectancy ≥ 3 months.
* Left Ventricular Ejection Fraction (LVEF)> 50% as assessed by MUGA scan or ECHO at screening.
* Normal pulmonary function with Force Vital Capacity (FVC) of at least 60% and DLCO of at least 50%.
* Adequate bone marrow, liver and renal function including the following:

  * Absolute neutrophil count ≥ 1.5 G/L, platelet count ≥ 100 G/L, and hemoglobin ≥ 10 g/dL)
  * AST/ALT ≤ 3 x upper limit of normal (ULN) (or ≤ 5.0 x ULN if liver metastasis) and total bilirubin ≤ 1.5 x ULN (≤ 2.5 x ULN if liver metastases),
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min according to Cockroft formula.
* Adequate contraceptive methods for the whole duration of the study and for up to 12 months after the last study drug administration.
* Mandatory affiliation with a health insurance company.
* Patients must provide written informed consent before any study specific procedures or assessments, and must be willing to comply with follow up assessments and procedures.

Exclusion Criteria:

* Chemotherapy within the last 2 weeks before inclusion; radiotherapy, or any other investigational agent within 14 days or 5 half-lives, whichever is longer prior to the first dose of study drug.
* Positive human anti-mouse antibody (HAMA) or human anti-chimeric antibody (HACA) response. HAMA/HACA assays will be performed only for patients previously treated by monoclonal antibodies.
* Uncontrolled arterial hypertension: systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg or both despite appropriate therapy.
* Patients with brain metastases.
* Previous history of high-dose chemotherapy with stem cell rescue.
* Chronic use of immunosuppressive drugs such as systemic corticosteroids.
* Previous therapy with monoclonal antibodies within 4 months before study entry.
* Clinically significant abnormal ECG (i.e. > grade 1) at inclusion.
* Prior history of other malignancies other than synovial sarcoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the subjects has been free of the disease for at least 3 years.
* No resolution of all specific toxicities (excluding alopecia) related to any prior anti-cancer therapy to Grade ≤ 1 according to the NCI CTCAE v4.
* Known immediate or delayed hypersensitivity reaction to 111In, 90Y, DTPA or any excipients of the investigational product.
* Psychological, familial, sociological, or geographical conditions that would limit compliance with study protocol requirements.
* Pregnant and breastfeeding women are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2015-02-03 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Part 1: Biodistribution and binding of OTSA101-DTPA-111In | 144 hours post-dose (dose administered at day -14)
  Limiting Event is defined as unacceptable/unexpected biodistribution/binding of the mAb, and/or absence of tumor uptake. Data review will be performed on a patient per patient basis. The Biodistribution and binding of OTSA101-DTPA-111In will be analyzed. The rate of Limiting Event will be summarized by a proportion together with its 95% confidence interval.
Part 2: Safety profile | During 1 year after randomization (day 0)
  The safety profile will be summarized with descriptive statistics including the following:
  * Occurrence of Severe Toxicities during the first 8 weeks post-injection of OTSA101-DTPA-90Y.
  * Occurrence of adverse events and serious adverse events during the study treatment period, including laboratory abnormalities, according to CTCAE v4.0 criteria.
  * Optimal recommended dose, defined as the dose level of OTSA101-DTPA-90Y with the best benefice-risk ratio taking into account the preliminary efficacy and safety data.

SECONDARY OUTCOMES:
Part 1: Pharmacokinetics parameters | They will be collected before the injection, (day -14) at 1, 2, 5, 24, 48, 72, 144 hours post dose and 7 days before randomisation
  The following PK parameters will be collected: Cmax, tmax, t½: terminal half-life; AUC, Cl, Vss: Volume of distribution. These PK parameters will be calculated using non-compartmental analysis.
Part 1: Safety profile of OTSA101-DTPA-111In | During 14 days
  The safety profile of OTSA101-DTPA-111In will be summarized with descriptive statistics. The occurrence of adverse events and serious adverse events during the whole imaging part, including laboratory abnormalities, will be summarized by a proportion together with its 95% confidence interval.
Part 2: Overall response rate | At 6 and 12 weeks after treatment
  The overall response rate is defined as the proportion of patients with a complete response or partial response on target lesions according to RECIST 1.1 criteria.
Part 2: Clinical benefit | At 6 and 12 weeks after treatment
  The clinical benefit rate is defined as the proportion of patients with a complete response or partial response or a stable disease on target lesions according to RECIST 1.1 criteria.
Part 2: Duration of response | At Week 6; Week12; Month 6; Month 9 and Month12 post Yttrium injection
  The duration of clinical response, measured from the time of first documented response until the first documented disease progression or death due to underlying cancer, will be described in responding subjects using descriptive statistics.
Part 2: Pharmacokinetics | They will be collected before the injection, (day 0) at 1, 5, 24, 48 hours post dose and 14, 28 days post dose and at the end of the study
  The following parameters will be collected: Cmax, tmax, t½: terminal half-life; AUC, Cl, Vss: Volume of distribution. Pharmacokinetics will be presented as descriptive statistics. Dose proportionality will be evaluated when applicable by an ANOVA mixed model. Accumulation will be assessed by Wilcoxon signed rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves BLAY, MD, PhD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France

REFERENCES:
- [Background] Jemal A, Siegel R, Xu J, Ward E. Cancer statistics, 2010. CA Cancer J Clin. 2010 Sep-Oct;60(5):277-300. doi: 10.3322/caac.20073. Epub 2010 Jul 7. PMID 20610543
- [Background] Clark MA, Fisher C, Judson I, Thomas JM. Soft-tissue sarcomas in adults. N Engl J Med. 2005 Aug 18;353(7):701-11. doi: 10.1056/NEJMra041866. No abstract available. PMID 16107623
- [Background] Ducimetiere F, Lurkin A, Ranchere-Vince D, Decouvelaere AV, Isaac S, Claret-Tournier C, Suignard Y, Salameire D, Cellier D, Alberti L, Bringuier PP, Blay JY, Ray-Coquard I. [Incidence rate, epidemiology of sarcoma and molecular biology. Preliminary results from EMS study in the Rhone-Alpes region]. Bull Cancer. 2010 Jun;97(6):629-41. doi: 10.1684/bdc.2010.1117. French. PMID 20504759
- [Background] Ladanyi M. Fusions of the SYT and SSX genes in synovial sarcoma. Oncogene. 2001 Sep 10;20(40):5755-62. doi: 10.1038/sj.onc.1204601. PMID 11607825
- [Background] Okcu MF, Munsell M, Treuner J, Mattke A, Pappo A, Cain A, Ferrari A, Casanova M, Ozkan A, Raney B. Synovial sarcoma of childhood and adolescence: a multicenter, multivariate analysis of outcome. J Clin Oncol. 2003 Apr 15;21(8):1602-11. doi: 10.1200/JCO.2003.07.008. PMID 12697886
- [Background] Trassard M, Le Doussal V, Hacene K, Terrier P, Ranchere D, Guillou L, Fiche M, Collin F, Vilain MO, Bertrand G, Jacquemier J, Sastre-Garau X, Bui NB, Bonichon F, Coindre JM. Prognostic factors in localized primary synovial sarcoma: a multicenter study of 128 adult patients. J Clin Oncol. 2001 Jan 15;19(2):525-34. doi: 10.1200/JCO.2001.19.2.525. PMID 11208847
- [Background] Laor T. MR imaging of soft tissue tumors and tumor-like lesions. Pediatr Radiol. 2004 Jan;34(1):24-37. doi: 10.1007/s00247-003-1086-3. Epub 2003 Dec 12. PMID 14673551
- [Background] Lewis JJ, Antonescu CR, Leung DH, Blumberg D, Healey JH, Woodruff JM, Brennan MF. Synovial sarcoma: a multivariate analysis of prognostic factors in 112 patients with primary localized tumors of the extremity. J Clin Oncol. 2000 May;18(10):2087-94. doi: 10.1200/JCO.2000.18.10.2087. PMID 10811674
- [Background] Singer S, Baldini EH, Demetri GD, Fletcher JA, Corson JM. Synovial sarcoma: prognostic significance of tumor size, margin of resection, and mitotic activity for survival. J Clin Oncol. 1996 Apr;14(4):1201-8. doi: 10.1200/JCO.1996.14.4.1201. PMID 8648375
- [Background] Adjuvant chemotherapy for localised resectable soft-tissue sarcoma of adults: meta-analysis of individual data. Sarcoma Meta-analysis Collaboration. Lancet. 1997 Dec 6;350(9092):1647-54. PMID 9400508
- [Background] Sleijfer S, Ouali M, van Glabbeke M, Krarup-Hansen A, Rodenhuis S, Le Cesne A, Hogendoorn PC, Verweij J, Blay JY. Prognostic and predictive factors for outcome to first-line ifosfamide-containing chemotherapy for adult patients with advanced soft tissue sarcomas: an exploratory, retrospective analysis on large series from the European Organization for Research and Treatment of Cancer-Soft Tissue and Bone Sarcoma Group (EORTC-STBSG). Eur J Cancer. 2010 Jan;46(1):72-83. doi: 10.1016/j.ejca.2009.09.022. PMID 19853437
- [Background] Le Cesne A, Blay JY, Judson I, Van Oosterom A, Verweij J, Radford J, Lorigan P, Rodenhuis S, Ray-Coquard I, Bonvalot S, Collin F, Jimeno J, Di Paola E, Van Glabbeke M, Nielsen OS. Phase II study of ET-743 in advanced soft tissue sarcomas: a European Organisation for the Research and Treatment of Cancer (EORTC) soft tissue and bone sarcoma group trial. J Clin Oncol. 2005 Jan 20;23(3):576-84. doi: 10.1200/JCO.2005.01.180. PMID 15659504
- [Background] Sleijfer S, Ray-Coquard I, Papai Z, Le Cesne A, Scurr M, Schoffski P, Collin F, Pandite L, Marreaud S, De Brauwer A, van Glabbeke M, Verweij J, Blay JY. Pazopanib, a multikinase angiogenesis inhibitor, in patients with relapsed or refractory advanced soft tissue sarcoma: a phase II study from the European organisation for research and treatment of cancer-soft tissue and bone sarcoma group (EORTC study 62043). J Clin Oncol. 2009 Jul 1;27(19):3126-32. doi: 10.1200/JCO.2008.21.3223. Epub 2009 May 18. PMID 19451427
- [Background] Fletcher CD. The evolving classification of soft tissue tumours: an update based on the new WHO classification. Histopathology. 2006 Jan;48(1):3-12. doi: 10.1111/j.1365-2559.2005.02284.x. PMID 16359532
- [Background] Lee YF, John M, Edwards S, Clark J, Flohr P, Maillard K, Edema M, Baker L, Mangham DC, Grimer R, Wooster R, Thomas JM, Fisher C, Judson I, Cooper CS. Molecular classification of synovial sarcomas, leiomyosarcomas and malignant fibrous histiocytomas by gene expression profiling. Br J Cancer. 2003 Feb 24;88(4):510-5. doi: 10.1038/sj.bjc.6600766. PMID 12592363
- [Background] Nielsen TO, West RB, Linn SC, Alter O, Knowling MA, O'Connell JX, Zhu S, Fero M, Sherlock G, Pollack JR, Brown PO, Botstein D, van de Rijn M. Molecular characterisation of soft tissue tumours: a gene expression study. Lancet. 2002 Apr 13;359(9314):1301-7. doi: 10.1016/S0140-6736(02)08270-3. PMID 11965276
- [Background] Allander SV, Illei PB, Chen Y, Antonescu CR, Bittner M, Ladanyi M, Meltzer PS. Expression profiling of synovial sarcoma by cDNA microarrays: association of ERBB2, IGFBP2, and ELF3 with epithelial differentiation. Am J Pathol. 2002 Nov;161(5):1587-95. doi: 10.1016/S0002-9440(10)64437-9. PMID 12414507
- [Background] Nagayama S, Katagiri T, Tsunoda T, Hosaka T, Nakashima Y, Araki N, Kusuzaki K, Nakayama T, Tsuboyama T, Nakamura T, Imamura M, Nakamura Y, Toguchida J. Genome-wide analysis of gene expression in synovial sarcomas using a cDNA microarray. Cancer Res. 2002 Oct 15;62(20):5859-66. PMID 12384549
- [Background] Ray-Coquard I, Le Cesne A, Whelan JS, Schoffski P, Bui BN, Verweij J, Marreaud S, van Glabbeke M, Hogendoorn P, Blay JY. A phase II study of gefitinib for patients with advanced HER-1 expressing synovial sarcoma refractory to doxorubicin-containing regimens. Oncologist. 2008 Apr;13(4):467-73. doi: 10.1634/theoncologist.2008-0065. PMID 18448563
- [Background] Koike J, Takagi A, Miwa T, Hirai M, Terada M, Katoh M. Molecular cloning of Frizzled-10, a novel member of the Frizzled gene family. Biochem Biophys Res Commun. 1999 Aug 19;262(1):39-43. doi: 10.1006/bbrc.1999.1161. PMID 10448064
- [Background] Hanaoka H, Katagiri T, Fukukawa C, Yoshioka H, Yamamoto S, Iida Y, Higuchi T, Oriuchi N, Paudyal B, Paudyal P, Nakamura Y, Endo K. Radioimmunotherapy of solid tumors targeting a cell-surface protein, FZD10: therapeutic efficacy largely depends on radiosensitivity. Ann Nucl Med. 2009 Jul;23(5):479-85. doi: 10.1007/s12149-009-0265-1. Epub 2009 May 2. PMID 19412654
- [Background] Nagayama S, Fukukawa C, Katagiri T, Okamoto T, Aoyama T, Oyaizu N, Imamura M, Toguchida J, Nakamura Y. Therapeutic potential of antibodies against FZD 10, a cell-surface protein, for synovial sarcomas. Oncogene. 2005 Sep 15;24(41):6201-12. doi: 10.1038/sj.onc.1208780. PMID 16007199
- [Background] Fukukawa C, Hanaoka H, Nagayama S, Tsunoda T, Toguchida J, Endo K, Nakamura Y, Katagiri T. Radioimmunotherapy of human synovial sarcoma using a monoclonal antibody against FZD10. Cancer Sci. 2008 Feb;99(2):432-40. doi: 10.1111/j.1349-7006.2007.00701.x. PMID 18271942
- [Background] Theuer CP, Leigh BR, Multani PS, Allen RS, Liang BC. Radioimmunotherapy of non-Hodgkin's lymphoma: clinical development of the Zevalin regimen. Biotechnol Annu Rev. 2004;10:265-95. doi: 10.1016/S1387-2656(04)10011-2. PMID 15504711
- [Background] Cheson BD. Radioimmunotherapy of non-Hodgkin lymphomas. Blood. 2003 Jan 15;101(2):391-8. doi: 10.1182/blood-2002-06-1793. Epub 2002 Sep 19. PMID 12393555
- [Background] Jain S, Xu R, Prieto VG, Lee P. Molecular classification of soft tissue sarcomas and its clinical applications. Int J Clin Exp Pathol. 2010 Apr 23;3(4):416-28. PMID 20490332
- [Background] Goldenberg DM. Advancing role of radiolabeled antibodies in the therapy of cancer. Cancer Immunol Immunother. 2003 May;52(5):281-96. doi: 10.1007/s00262-002-0348-5. Epub 2003 Mar 11. PMID 12700944
- [Background] Verhaar-Langereis MJ, Zonnenberg BA, de Klerk JM, Blijham GH. Radioimmunodiagnosis and therapy. Cancer Treat Rev. 2000 Feb;26(1):3-10. doi: 10.1053/ctrv.1999.0146. PMID 10660488
- [Background] Pinkas L, Robins PD, Forstrom LA, Mahoney DW, Mullan BP. Clinical experience with radiolabelled monoclonal antibodies in the detection of colorectal and ovarian carcinoma recurrence and review of the literature. Nucl Med Commun. 1999 Aug;20(8):689-96. doi: 10.1097/00006231-199908000-00002. PMID 10451876
- [Background] Sodee DB, Malguria N, Faulhaber P, Resnick MI, Albert J, Bakale G. Multicenter ProstaScint imaging findings in 2154 patients with prostate cancer. The ProstaScint Imaging Centers. Urology. 2000 Dec 20;56(6):988-93. doi: 10.1016/s0090-4295(00)00824-4. PMID 11113745
- [Background] Tsai SW, Sun Y, Williams LE, Raubitschek AA, Wu AM, Shively JE. Biodistribution and radioimmunotherapy of human breast cancer xenografts with radiometal-labeled DOTA conjugated anti-HER2/neu antibody 4D5. Bioconjug Chem. 2000 May-Jun;11(3):327-34. doi: 10.1021/bc9901292. PMID 10821648
- [Background] Milowsky MI, Nanus DM, Kostakoglu L, Vallabhajosula S, Goldsmith SJ, Bander NH. Phase I trial of yttrium-90-labeled anti-prostate-specific membrane antigen monoclonal antibody J591 for androgen-independent prostate cancer. J Clin Oncol. 2004 Jul 1;22(13):2522-31. doi: 10.1200/JCO.2004.09.154. Epub 2004 Jun 1. PMID 15173215
- [Background] Tempero M, Leichner P, Baranowska-Kortylewicz J, Harrison K, Augustine S, Schlom J, Anderson J, Wisecarver J, Colcher D. High-dose therapy with 90Yttrium-labeled monoclonal antibody CC49: a phase I trial. Clin Cancer Res. 2000 Aug;6(8):3095-102. PMID 10955789
- [Background] Richman CM, DeNardo SJ, O'Donnell RT, Goldstein DS, Shen S, Kukis DL, Kroger LA, Yuan A, Boniface GR, Griffith IJ, DeNardo GL. Dosimetry-based therapy in metastatic breast cancer patients using 90Y monoclonal antibody 170H.82 with autologous stem cell support and cyclosporin A. Clin Cancer Res. 1999 Oct;5(10 Suppl):3243s-3248s. PMID 10541370
- [Background] Pai-Scherf LH, Carrasquillo JA, Paik C, Gansow O, Whatley M, Pearson D, Webber K, Hamilton M, Allegra C, Brechbiel M, Willingham MC, Pastan I. Imaging and phase I study of 111In- and 90Y-labeled anti-LewisY monoclonal antibody B3. Clin Cancer Res. 2000 May;6(5):1720-30. PMID 10815890
- [Background] Pless M, Waldherr C, Maecke H, Buitrago C, Herrmann R, Mueller-Brand J. Targeted radiotherapy for small cell lung cancer using 90Yttrium-DOTATOC, an Yttrium-labelled somatostatin analogue: a pilot trial. Lung Cancer. 2004 Sep;45(3):365-71. doi: 10.1016/j.lungcan.2004.02.020. PMID 15301877
- [Background] Forrer F, Riedweg I, Maecke HR, Mueller-Brand J. Radiolabeled DOTATOC in patients with advanced paraganglioma and pheochromocytoma. Q J Nucl Med Mol Imaging. 2008 Dec;52(4):334-40. Epub 2008 May 16. PMID 18480742
- [Background] Tubiana M, Koscielny S. On clonogenic tumour cells and metastasis-forming cells. Nat Rev Cancer. 2008 Dec;8(12):990; author reply 990. doi: 10.1038/nrc2419-c1. No abstract available. PMID 19029960
- [Background] Betts AM, Clark TH, Yang J, Treadway JL, Li M, Giovanelli MA, Abdiche Y, Stone DM, Paralkar VM. The application of target information and preclinical pharmacokinetic/pharmacodynamic modeling in predicting clinical doses of a Dickkopf-1 antibody for osteoporosis. J Pharmacol Exp Ther. 2010 Apr;333(1):2-13. doi: 10.1124/jpet.109.164129. Epub 2010 Jan 20. PMID 20089807
- [Background] Leveque D, Wisniewski S, Jehl F. Pharmacokinetics of therapeutic monoclonal antibodies used in oncology. Anticancer Res. 2005 May-Jun;25(3c):2327-43. PMID 16080460
- [Background] Kelly MP, Lee FT, Smyth FE, Brechbiel MW, Scott AM. Enhanced efficacy of 90Y-radiolabeled anti-Lewis Y humanized monoclonal antibody hu3S193 and paclitaxel combined-modality radioimmunotherapy in a breast cancer model. J Nucl Med. 2006 Apr;47(4):716-25. PMID 16595507
- [Background] Knox SJ, Goris ML, Trisler K, Negrin R, Davis T, Liles TM, Grillo-Lopez A, Chinn P, Varns C, Ning SC, Fowler S, Deb N, Becker M, Marquez C, Levy R. Yttrium-90-labeled anti-CD20 monoclonal antibody therapy of recurrent B-cell lymphoma. Clin Cancer Res. 1996 Mar;2(3):457-70. PMID 9816191
- [Background] Nademanee A, Forman S, Molina A, Fung H, Smith D, Dagis A, Kwok C, Yamauchi D, Anderson AL, Falk P, Krishnan A, Kirschbaum M, Kogut N, Nakamura R, O'donnell M, Parker P, Popplewell L, Pullarkat V, Rodriguez R, Sahebi F, Smith E, Snyder D, Stein A, Spielberger R, Zain J, White C, Raubitschek A. A phase 1/2 trial of high-dose yttrium-90-ibritumomab tiuxetan in combination with high-dose etoposide and cyclophosphamide followed by autologous stem cell transplantation in patients with poor-risk or relapsed non-Hodgkin lymphoma. Blood. 2005 Oct 15;106(8):2896-902. doi: 10.1182/blood-2005-03-1310. Epub 2005 Jul 7. PMID 16002426
- [Background] Lhommel R, van Elmbt L, Goffette P, Van den Eynde M, Jamar F, Pauwels S, Walrand S. Feasibility of 90Y TOF PET-based dosimetry in liver metastasis therapy using SIR-Spheres. Eur J Nucl Med Mol Imaging. 2010 Aug;37(9):1654-62. doi: 10.1007/s00259-010-1470-9. Epub 2010 Apr 27. PMID 20422185
- [Background] Baechler S, Hobbs RF, Jacene HA, Bochud FO, Wahl RL, Sgouros G. Predicting hematologic toxicity in patients undergoing radioimmunotherapy with 90Y-ibritumomab tiuxetan or 131I-tositumomab. J Nucl Med. 2010 Dec;51(12):1878-84. doi: 10.2967/jnumed.110.079947. PMID 21098795
- [Background] Minarik D, Sjogreen-Gleisner K, Linden O, Wingardh K, Tennvall J, Strand SE, Ljungberg M. 90Y Bremsstrahlung imaging for absorbed-dose assessment in high-dose radioimmunotherapy. J Nucl Med. 2010 Dec;51(12):1974-8. doi: 10.2967/jnumed.110.079897. Epub 2010 Nov 15. PMID 21078799
- [Background] Rault E, Staelens S, Van Holen R, De Beenhouwer J, Vandenberghe S. Fast simulation of yttrium-90 bremsstrahlung photons with GATE. Med Phys. 2010 Jun;37(6):2943-50. doi: 10.1118/1.3431998. PMID 20632606
- [Background] Walrand S, Flux GD, Konijnenberg MW, Valkema R, Krenning EP, Lhommel R, Pauwels S, Jamar F. Dosimetry of yttrium-labelled radiopharmaceuticals for internal therapy: 86Y or 90Y imaging? Eur J Nucl Med Mol Imaging. 2011 May;38 Suppl 1:S57-68. doi: 10.1007/s00259-011-1771-7. Epub 2011 Mar 11. PMID 21484382
- [Background] Shen D, Fritz T, Wu GL, Kulik B, Palestrant D, Unger E. Block co-polymeric magnetic resonance contrast agents. Invest Radiol. 1994 Jun;29 Suppl 2:S217-9. doi: 10.1097/00004424-199406001-00072. No abstract available. PMID 7928236
- [Derived] Giraudet AL, Cassier PA, Iwao-Fukukawa C, Garin G, Badel JN, Kryza D, Chabaud S, Gilles-Afchain L, Clapisson G, Desuzinges C, Sarrut D, Halty A, Italiano A, Mori M, Tsunoda T, Katagiri T, Nakamura Y, Alberti L, Cropet C, Baconnier S, Berge-Montamat S, Perol D, Blay JY. A first-in-human study investigating biodistribution, safety and recommended dose of a new radiolabeled MAb targeting FZD10 in metastatic synovial sarcoma patients. BMC Cancer. 2018 Jun 8;18(1):646. doi: 10.1186/s12885-018-4544-x. PMID 29884132